CLINICAL TRIAL: NCT03830905
Title: Double-blind Randomized Placebo-controlled Comparative Multicenter Study to Assess the Safety, Tolerability and Efficacy of XC221 in a Dose of 200mg Per Day in Patients With Uncomplicated Influenza or Other ARVI
Brief Title: Study to Assess Efficacy and Safety of XC221 200 mg in the Treatment of Influenza or Other ARVI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PHARMENTERPRISES LLC (Industry)
Collaborators: RSV Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARI-XC221-03
Record Dates: First submitted 2019-01-30; First posted 2019-02-05 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Influenza; Acute Respiratory Viral Infections
MeSH Terms: conditions — Influenza, Human | interventions — XC221

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XC221 (Experimental): XC221 200 mg orally. 2 tablets of XC221 100 mg once daily during 3 days of treatment period
  Interventions: Drug: XC221
- Placebo (Placebo Comparator): Placebo orally. 2 tablets of Placebo once daily during 3 days of treatment period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC221 — Participants will receive 200 mg XC221 once a day during 3 days
  Arms: XC221
Drug: Placebo — Participants will receive Placebo once a day during 3 days
  Arms: Placebo

SUMMARY:
The innovative drug XC221 is planned for use in treatment of acute respiratory viral infections in a double-blind, randomized, placebo-controlled, comparative multicenter study assessing the safety, tolerability and efficacy of XC221 at a dose of 200 mg per day in patients with uncomplicated influenza or other acute respiratory viral infections during the 3-days treatment.

DETAILED DESCRIPTION:
A double-blind, randomized, placebo-controlled, comparative multicenter study in two groups. A total of 120 patients with uncomplicated influenza or other acute respiratory viral infections are planned to be randomized. Patients will be randomized into 2 groups: 60 patients in the treatment group 200 mg XC221 and 60 patients in the placebo group. The purpose of the clinical trial is to assess the safety, tolerability and efficacy of the drug XC21 in treatment of influenza or other acute respiratory viral infections. The primary objective is to demonstrate the difference between the groups in the time of the onset of sustained improvement in clinical symptoms according to the Modified Jackson Scale. The study will consist of the following periods: screening (duration not more than 36 hours from the moment of the first symptoms of the disease), treatment period (3 days), follow-up period (11 ± 1 days after completion of treatment with the study drug/placebo). The duration of participation in the study for each patient is no more than 16 days and 12 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes aged 18 years and older.
2. Clinically diagnosed influenza or ARVI mild or moderate severity.
3. Patient's body temperature ≥37.5ºС and at least 1 symptom from Modified Jackson Scale estimated more than 2 points.
4. Uncomplicated course of influenza or ARVI based on clinical estimations.
5. The first 36 hours from the beginning of symptoms of influenza or ARVI.
6. Women of reproductive age (who are not in menopause and who have not undergone surgical sterilization) and men who have sexual activity should use a reliable method of contraception (acceptable methods of contraception in this study are: intrauterine devices, oral contraceptives, contraceptive patch, long-acting injectable contraceptives, a double barrier method (condom and diaphragm with spermicide) throughout the study period.
7. Compliance with the treatment regimen, visits and laboratory examinations provided by the protocol.
8. Signed Informed Consent Form.

Exclusion Criteria:

1. Complications of influenza or ARVI (including the presence / development of bacterial infection).
2. The need for inpatient treatment of influenza and ARVI.
3. Hypersensitivity to excipients of the drug XC221 or placebo.
4. Antiviral medications 7 days prior to screening (antiviral agents, interferons and interferon inducers, drugs that have immunomodulating action) or anti-infective agents of systemic or local action.
5. Severe infection with signs of cardiovascular insufficiency development and other manifestations of infectious-toxic shock, as well as with the presence of neuroinfection syndrome (encephalic and meningoencephalic reactions, polyradiculoneuritis, neuritis).
6. Signs of of viral pneumonia symptoms (the presence of two or more of the following symptoms): dyspnea, chest pain when coughing, systemic cyanosis, dullness of percussion sound with a symmetrical evaluation of the upper and lower sections of the lungs).
7. Infectious diseases during the last week before including into the study.
8. Bronchial asthma, COPD, pulmonary emphysema in history.
9. History of increased convulsive activity.
10. Severe, decompensated or unstable somatic diseases (any diseases or conditions that are life-threatening or may worsen the patient's prognosis, and make him/her ineligible for the clinical study).
11. History of oncological diseases, HIV, tuberculosis.
12. Drug or alcohol abuse.
13. Lactose intolerance, lactase deficiency, glucose-galactose malabsorption.
14. Participation in any other clinical trial in the last 90 days.
15. Pregnancy or lactation.
16. Military or prison populations.
17. Impossibility or inability to comply with the study procedures.
18. A member of the investigator's family or other person interested in the results of the study.
19. Deviations from laboratory standards, which prevent the inclusion of the patient in the study according to the Investigator.
20. A history of kidney failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Time to sustained improvement in clinical symptoms according to the Modified Jackson Scale for measuring respiratory symptoms. | From the moment of the first dose up to Day 14
  The time before the onset of sustained improvement in clinical symptoms according to the Modified Jackson Scale (no more than 1 point for each symptom), measured in hours from the moment of the first dose of the drug.
  Modified Jackson Scale measures individuals' subjective ratings the severity of 12 respiratory symptoms. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 32 points) is a sum of the point for each symptom.

SECONDARY OUTCOMES:
The time before the onset of persistent improvement in clinical symptoms according to the Modified Jackson Scale for measuring respiratory symptoms (0 points). | From the moment of the first dose up to Day 14
  The time of the first assessment of 3 consecutive ratings on the Modified Jackson Scale, in which all the clinical symptoms were 0 points.
  Modified Jackson Scale measures individuals' subjective ratings the severity of 12 respiratory symptoms. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 32 points) is a sum of the point for each symptom.
The time before the onset of persistent improvement in clinical symptoms according to the Modified Jackson Scale for measuring respiratory symptoms. | From the moment of the first dose up to Day 14
  Total score of no more than 3 points, when there is no more than 1 point for each symptom, measured in hours from the moment of taking the first dose of the drug.
  Modified Jackson Scale measures individuals' subjective ratings the severity of 12 respiratory symptoms. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 32 points) is a sum of the point for each symptom.
Time to normalization of body temperature. | From the moment of the first dose up to Day 14
  Measured in hours. Normalization means the establishment of body temperature below 37° C without a rise above these values in the subsequent observation period.
The average score according to the Modified Jackson Scale for measuring respiratory symptoms at the 1st, 2nd, 3rd, 4th, 5th, 6th, 7th, 8th days. | From the moment of the first dose up to Day 14
  The average score according to the Modified Jackson Scale on the 1st, 2nd, 3rd, 4th, 5th, 6th, 7th, 8th days.
  Modified Jackson Scale measures individuals' subjective ratings the severity of 12 respiratory symptoms. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 32 points) is a sum of the point for each symptom.
The proportion of patients with a sum of not more than 3 points according to the Modified Jackson Scale for measuring respiratory symptoms at the 1st, 2nd, 3rd, 4th, 5th, 6th , The 7th, 8th days | From the moment of the first dose up to Day 14
  Score for each symptom should be no higher than 1 point at the 1st, 2nd, 3rd, 4th, 5th, 6th , The 7th, 8th days from the moment of the start of treatment.
  Modified Jackson Scale measures individuals' subjective ratings the severity of 12 respiratory symptoms. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 32 points) is a sum of the point for each symptom.
The proportion of patients with the normalization of body temperature on the first - the 14th days from the start of treatment; | From the moment of the first dose up to Day 14
Time to disappearance (0 points) of each of the symptoms according to the Modified Jackson Scale for measuring respiratory symptoms. | From the moment of the first dose up to Day 14
  Symptom (sneezing, rhinorrhea, nasal congestion, cough, fever, malaise, chills, headache, myalgia, sore throat, tickling, hoarseness) manifested at the level of 2 or 3 points at the first assessment at Visit 0 (Day 0).
  Modified Jackson Scale measures individuals' subjective ratings the severity of 12 respiratory symptoms. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 32 points) is a sum of the point for each symptom.
The proportion of patients with 0 points score for each of the symptoms according to the Modified Jackson Scale for measuring respiratory symptoms. | From the moment of the first dose up to Day 14
  Modified Jackson Scale (sneezing, rhinorrhea, nasal congestion, cough, fever, malaise, chills, headache, myalgia, sore throat, tickling, hoarseness) at the 2nd, 3rd 2nd, 4th, 5th, 6th, 7th and 8th days from the moment of the start of treatment in a population of patients with the corresponding symptom shown at the level of 2 or 3 points at Visit 0 (Day 0).
  Modified Jackson Scale measures individuals' subjective ratings the severity of 12 respiratory symptoms. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 32 points) is a sum of the point for each symptom.
The proportion of patients with a detected viral pathogen | From the moment of the first dose up to Day 14
  The proportion of patients with a detected viral pathogen at Visit 0, Visit 4 and Visit 6.
The proportion of patients with a detected viral pathogen at Visit 4 and Visit 6 compared with the initial proportion of such patients in the XC221. | From the moment of the first dose up to Day 14
The frequency of adverse events (AEs) and serious adverse events (SAEs) in the XC221 treatment group and in the placebo group. | From the moment of the first dose up to Day 14

OTHER OUTCOMES:
The average concentration of MxA protein in the blood at Visit 1, Visit 4 and at Visit 6. | From Day 1 up to Day 6
Changes in the concentration of MxA protein in the blood at Visit 4 and at Visit 6 compared to Visit 1. | From Day 1 up to Day 6
The average concentration of C-reactive protein in the blood at Visit 1, Visit 4 and Visit 6. | From Day 1 up to Day 6
Changes in the concentration of C-reactive protein in the blood at Visit 4 and Visit 6 compared to Visit 1. | From Day 1 up to Day 6
The average concentration of cytokines at Visit 1, Visit 4 and at Visit 6. | From Day 1 up to Day 6
  The average concentration of 6Ckine, BCA-1, CTACK, ENA-78, Eotaxin, Eotaxin-2, Eotaxin-3, Fractalkine, GCP-2, GM-CSF, Gro-α, Gro-β, I-309, IFN- γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-16, IP-10, I-TAC, MCP-1, MCP-2, MCP-3, MCP-4, MDC, MIF, MIG, MIP-1α, MIP-1δ, MIP-3α, MIP-3β, MPIF-1, SCYB16, SDF-1α + β, TARC, TECK, TNF-α in blood at Visit 1, Visit 4 and at Visit 6.
The percentage change in the concentration of cytokines at Visit 4 and at Visit 6 compared with Visit 1. | From Day 1 up to Day 6
  The percentage change in the concentration of 6Ckine, BCA-1, CTACK, ENA-78, Eotaxin, Eotaxin-2, Eotaxin-3, Fractalkine, GCP-2, GM-CSF, Gro-α, Gro-β, I-309, IFN -γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-16, IP-10, I-TAC, MCP-1, MCP-2, MCP-3 , MCP-4, MDC, MIF, MIG, MIP-1α, MIP-1δ, MIP-3α, MIP-3β, MPIF-1, SCYB16, SDF-1α + β, TARC, TECK, TNF-α in blood at Visit 4 and Visit 6 compared with Visit 1.
Correlation between the concentration of cytokines/chemokines and the assessment of the Modified Jackson scale for measuring respiratory symptoms (in dynamics). | From the moment of the first dose up to Day 14
  Modified Jackson Scale measures individuals' subjective ratings the severity of 12 respiratory symptoms. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 32 points) is a sum of the point for each symptom.
The average concentration of cytokines in a smear from the mucosa of the nasopharynx and oropharyngeal at Visit 1, Visit 4 and Visit 6 | From Day 1 up to Day 6
  The average concentration of 6Ckine, BCA-1, CTACK, ENA-78, Eotaxin, Eotaxin-2, Eotaxin-3, Fractalkine, GCP-2, GM-CSF, Gro-α, Gro-β, I-309, IFN- γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-16, IP-10, I-TAC, MCP-1, MCP-2, MCP-3, MCP-4, MDC, MIF, MIG, MIP-1α, MIP-1δ, MIP-3α, MIP-3β, MPIF-1, SCYB16, SDF-1α + β, TARC, TECK, TNF-α in a smear from the mucosa of the nasopharynx and oropharyngeal at Visit 1, Visit 4 and Visit 6.
The percentage change in the concentration of cytokines in a smear from the mucous membrane of the nasopharynx and oropharynx of patients on Visit 4 and on Visit 6 compared to Visit 1. | From Day 1 up to Day 6
  The percentage change in the concentration of 6Ckine, BCA-1, CTACK, ENA-78, Eotaxin, Eotaxin-2, Eotaxin-3, Fractalkine, GCP-2, GM-CSF, Gro-α, Gro-β, I-309, IFN- γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-16, IP-10, I-TAC, MCP-1, MCP-2, MCP-3, MCP-4, MDC, MIF, MIG, MIP-1α, MIP-1δ, MIP-3α, MIP-3β, MPIF-1, SCYB16, SDF-1α + β, TARC, TECK, TNF-α in a smear from the mucous membrane of the nasopharynx and oropharynx of patients on Visit 4 and on Visit 6 compared to Visit 1.

CONTACTS AND LOCATIONS:
Locations (16):
- Russia (16):
  - Federal State Budgetary Institution of Health "Northern Medical Clinical Center named after NA Semashko of the Federal Medical and Biological Agency", Arkhangelsk
  - Regional State Budgetary Institution of Health "Belgorod Regional Clinical Hospital of St. Joasaph", Belgorod
  - City Clinical Hospital №9, Izhevsk
  - Kuban State Medical University, Krasnodar
  - State budget institution of health care of the Moscow region "Krasnogorsk city hospital number 1", Krasnogorsk
  - Non-governmental Healthcare Institution "N.A.Semashko Road Clinical Hospital at the Lyublino station of the open joint-stock company "Russian Railways", Moscow
  - Federal State Budgetary Educational Institution of Higher Education "Ryazan State Medical University named after Academician I.P. Pavlova" of the Ministry of Health of the Russian Federation, Ryazan
  - Ryazan State Medical University n.a. Pavlov, Ryazan
  - The Center for Prevention and Fight about AIDS and Infectious Diseases, Saint Petersburg
  - LLC "Aurora Medi", Saint Petersburg
  - The Consulting and Diagnostic Center with out-patient help of the Administration of the President of the Russian Federation, Saint Petersburg
  - Research Institute of Influenza, Saint Petersburg
  - City Clinical Hospital №40 of Kurortny District, Saint Petersburg
  - LLC "Astarta", Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "Yaroslavl State Medical University" of the Ministry of Health of the Russian Federation, Yaroslavl
  - State Budgetary Healthcare Institution (SBHI) of Yaroslavl region, Yaroslavl

IPD SHARING:
Plan to Share IPD: No